CLINICAL TRIAL: NCT02339922
Title: A Window Study of Ixazomib in Untreated Indolent B-NHL
Brief Title: Ixazomib Citrate and Rituximab in Treating Patients With Indolent B-cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9571; NCI-2016-00401 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9224; 9571 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1716009 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-12-30; First posted 2015-01-16 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Recurrent Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Refractory Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — ixazomib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (ixazomib citrate, rituximab) (Experimental): Patients receive ixazomib citrate orally (PO) on days 1, 8 ,15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Upon completion of 6 cycles of ixazomib citrate therapy, patients also receive rituximab intravenously (IV) once weekly for 4 doses total, followed by ixazomib citrate alone, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83; Rituximab Biosimilar SIBP-02

SUMMARY:
This phase II trial studies how well ixazomib citrate and rituximab work in treating patients with B-cell non-Hodgkin lymphoma that grows slowly (indolent). Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving ixazomib citrate together with rituximab may work better in treating indolent B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive ixazomib citrate orally (PO) on days 1, 8 ,15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Upon completion of 6 cycles of ixazomib citrate therapy, patients also receive rituximab intravenously (IV) once weekly for 4 doses total, followed by ixazomib citrate alone, until disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Patients must have a diagnosis of one of the following B-NHL malignancies: chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), or Waldenstrom macroglobulinemia (WM)/ lymphoplasmacytic lymphoma (LPL); patients with mucosa associated lymphoid tissue (MALT) subtype of MZL may have relapsed or refractory disease after a course of antibiotic therapy; otherwise, patients will not have received standard systemic treatment for their B-NHL before the time of study enrollment; standard systemic therapy is defined by including any of the following agents, representing a comprehensive list of recommended front-line agents used in the treatment of B-NHL: cytotoxic chemotherapies (bendamustine, cyclophosphamide, doxorubicin, vincristine, chlorambucil, cytarabine, gemcitabine, platinum drugs, etoposide); anti-CD20 antibodies (obinutuzumab, ofatumumab, rituximab); lenalidomide; ibritumomab tiuxetan; proteasome inhibitors (bortezomib, carfilzomib); tyrosine kinase inhibitors (ibrutinib, acalabrutinib, idelalisib); alemtuzumab; corticosteroids unless given for an indication other than treating the B-NHL; or other therapy as determined by the principal investigator (PI)

  * Disease: CLL/SLL; Criteria for diagnosis: histopathologic or flow cytometric confirmation
  * Disease: FL; Criteria for diagnosis: histopathologic confirmation
  * Disease: MZL; Criteria for diagnosis: histopathologic confirmation
  * Disease: MCL; Criteria for diagnosis: histopathologic confirmation
  * Disease: WM/LPL; Criteria for diagnosis: Per World Health Organization (WHO) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3 or >= 500/mm^3 if neutropenia is attributed to B-NHL (involvement of bone marrow) without growth factor support
* Platelet count >= 100,000/mm^3 or >= 75,000/mm^3 if thrombocytopenia is attributed to B-NHL (involvement of bone marrow or due to splenomegaly or immune thrombocytopenic purpura); platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30 mL/min
* Patients are required to meet criteria for initiation of therapy for their B-NHL according to published guidelines by the National Comprehensive Cancer Network (NCCN)
* Patients must have measurable disease defined by at least one of the following criteria:

  * Lesions greater than 1.5 cm that can be accurately measured in two dimensions by computed tomography (CT) (preferred), or magnetic resonance imaging (MRI), and are not included in any prior field of radiation given to treat B-NHL
  * In patients with CLL, circulating lymphocytes >= 5,000 / mm^3
  * In patients with WM/LPL, measurable serum monoclonal immunoglobulin M (IgM)

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Major surgery within 14 days before enrollment
* Known central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, cardiac arrhythmias, or congestive heart failure, and unstable angina or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of ginkgo biloba or St. John's wort
* Known ongoing or known active systemic infection, known active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to ixazomib, its analogues, or excipients in the various formulations of ixazomib
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed (> 2 years before study enrollment) with another malignancy and have any evidence of residual disease that is symptomatic or requiring treatment; (this may be waived at the discretion of the principal investigator for patients in complete remission if they have not received systemic therapy); patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 2 peripheral neuropathy, or grade 1 with pain on clinical examination during the screening period
* Participation in other clinical trials with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial
* Patients may not have impending organ compromise from disease as assessed by their treating physician
* Prior treatment of B-NHL with radiation therapy, non-standard systemic therapy, or antibiotics (in cases of MZL) within 21 days of the first dose of ixazomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2031-01-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (complete response [CR] + partial response [PR]) in patients with chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), follicular lymphoma (FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL) | Up to 5 years
  ORR will be calculated for all treated patients for each disease cohort. The corresponding 95% two-sided confidence interval will be derived.
ORR (CR + very good PR + PR + minor response) in patients with Waldenstrom macroglobulinemia (WM)/ lymphoplasmacytic lymphoma (LPL) | Up to 5 years
  ORR will be calculated for all treated patients for each disease cohort. The corresponding 95% two-sided confidence interval will be derived.

SECONDARY OUTCOMES:
Duration of response (DOR) | From the time by which the measurement criteria are met for CR or PR, whichever is recorded first, until death or the first date by which recurrent or progressive disease is objectively documented, assessed up to 5 years
  DOR will be calculated to determine durability. Non-responders will be excluded from the analysis of DOR. Kaplan Meier methodology will be used to estimate event-free curves.
Progression-free survival (PFS) | Time from the first study drug administration to the first occurrence of lymphoma progression or death from any cause, assessed up to 5 years
  Data for subjects without disease progression or death will be censored at the date of the last tumor assessment. Kaplan-Meier methodology will be used to estimate the event-free curves.
Overall survival | Up to 5 years
CR rate | Up to 5 years
Time to next therapy (TNT) | From the time of first study drug administration until the date of subsequent the first subsequent therapy given to treat the B-NHL, assessed up to 5 years
  Data for subjects that have not received additional anti-neoplastic therapy will be censored at the date of last known contact.
Incidence of adverse events (AEs) | Up to 30 days after administration of the last dose of ixazomib citrate
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Safety summaries will include tabulations in the form of tables. The frequency of treatment-emergent AE's will be summarized. Additional AE summaries will include AE frequency by AE severity and relationship to the study drug. AE's requiring discontinuation of the study drug will be summarized separately, both overall and by AE severity and by relationship to the study drug. Clinically significant abnormal laboratory values will be summarized over study visits.

OTHER OUTCOMES:
Identification of clinical features (i.e. Mantle Cell International Prognostic score, Follicular Lymphoma International Prognostic Index score, and International Prognostic Scoring System score) and biomarker expression levels | Up to 5 years
Single nucleotide profile (SNP) genotyping for PSMB1 P11A | Up to 5 years
  SNP genotyping for PSMB1 P11A will be performed and will be correlated with response to ixazomib citrate and ixazomib citrate plus rituximab.
Gene expression profiling on tumor specimens | Up to 5 years
  Will be correlated with response to rituximab.
Tumor expression of cluster of differentiation 68, nuclear transcription factor kappa-B, p65, p27, and proteasome subunit, alpha-type, 5 by immunohistochemistry | Up to 5 years
  Will be correlated with response to ixazomib citrate and ixazomib citrate plus rituximab.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graf SA, Lynch RC, Ujjani CS, Gooley TA, Rasmussen H, Coffey DG, Cowan AJ, Smith SD, Shadman M, Warren EH, Libby EN, Greninger AL, Fromm JR, Gopal AK. Efficacy, safety, and molecular response predictors of oral ixazomib and short-course rituximab in untreated iNHL. Blood Adv. 2023 Mar 14;7(5):687-696. doi: 10.1182/bloodadvances.2022008628. PMID 36385536